CLINICAL TRIAL: NCT00866736
Title: A Phase II Study of Dasatinib in Patients With Imatinib Resistant or Intolerant Chronic Myeloid Leukemia
Brief Title: A Study of Dasatinib in Patients With Imatinib Resistant or Intolerant Chronic Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kanto CML Study Group (Other)
Collaborators: Epidemiological and Clinical Research Information Network (Other)
Responsible Party: Hisashi Sakamaki, Tokyo Metropolitan Cancer and Infectious diseases Center Komagome Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KCSG-01
Record Dates: First submitted 2009-03-18; First posted 2009-03-20 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2010-12

CONDITIONS: Chronic Myeloid Leukemia
Keywords: chronic myeloid leukemia; dasatinib; chronic phase myeloid leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Chronic-Phase | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- dasatinib (Experimental)
  Interventions: Drug: dasatinib

INTERVENTIONS:
Drug: dasatinib — 100mg QD
  Other Names: BMS-354825

SUMMARY:
The purpose of this study is to evaluate the efficacy and the safety of dasatinib in subject with chronic phase chronic myeloid leukemia(CML) who are either resistant to or intolerant of imatinib mesylate.

ELIGIBILITY:
Inclusion Criteria:

* Signed Written Informed Consent
* Subjects with chronic phase chronic myeloid leukemia (CML)
* Subjects resistant/intolerant to imatinib
* Subjects presenting:

  1. ECOG performance status (PS) score 0-2
  2. Adequate hepatic function
  3. Adequate renal function
  4. Adequate lung function

Exclusion Criteria:

* Concurrent malignancy other than CML
* Women who are pregnant or breastfeeding
* Concurrent pleural effusion
* Uncontrolled or significant cardiovascular disease
* A serious uncontrolled medical disorder that would impair the ability of the subjects to receive protocol therapy.
* Prior therapy with dasatinib
* Subjects with T315I and/or F317L BCR-ABL point mutations

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2009-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
rate of Major Molecular Responses (MMR) in chronic phase chronic myeloid leukemia subjects | at 12 months

SECONDARY OUTCOMES:
safety after treatment with dasatinib | 2 year
rate of Complete Cytogenetic Response(CCyR) | 2 year
rate of Complete Hematologic Response (CHR) | 2 year
efficacy on patients with BCR-ABL point mutations | 2 year
progression free survival | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Hisashi Sakamaki, MD.PhD, Principal Investigator — Tokyo Metropolitan Cancer and Infectious diseases Center Komagome Hospital
Locations (1):
- Tokyo Metropolitan Cancer and Infectious diseases Center Komagome Hospital, Bunkyo-ku, Tokyo, Japan

REFERENCES:
- [Derived] Inokuchi K, Kumagai T, Matsuki E, Ohashi K, Shinagawa A, Hatta Y, Takeuchi J, Yoshida C, Wakita H, Kozai Y, Shirasugi Y, Fujisawa S, Iwase O, Yano S, Okamoto S, Oba K, Sakamoto J, Sakamaki H. Efficacy of molecular response at 1 or 3 months after the initiation of dasatinib treatment can predict an improved response to dasatinib in imatinib-resistant or imatinib-intolerant Japanese patients with chronic myelogenous leukemia during the chronic phase. J Clin Exp Hematop. 2014;54(3):197-204. doi: 10.3960/jslrt.54.197. PMID 25501110